CLINICAL TRIAL: NCT03238430
Title: Management of Pain Post Hepatectomy : Infiltration of Local Anesthetics Versus Continuous Spinal Analgesia .
Acronym: CATHEPAT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013_48; 2014-003317-28 (EudraCT Number)
Record Dates: First submitted 2017-07-31; First posted 2017-08-03 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2020-08

CONDITIONS: Pain, Postoperative
Keywords: Intrathecal morphine, continuous wound infiltration
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ropivacaine infiltration (Experimental): Continuous infiltration of local anesthetics + PCA morphine.
  Interventions: Drug: intrathecal morphine; Drug: Morphine PCA
- intrathecal morphine (Experimental): Rachianalgesia + PCA morphine
  Interventions: Drug: Morphine PCA; Drug: Ropivacaine infiltration
- morphine PCA (Active Comparator): PCA morphine alone
  Interventions: Drug: Morphine PCA

INTERVENTIONS:
Drug: intrathecal morphine — A single intrathecal injection of 300 micrograms of Morphine preoperatively, just before induction.
  Arms: Ropivacaine infiltration
Drug: Morphine PCA — a postoperative Morphine PCA
Drug: Ropivacaine infiltration — Ropivacaine 2mg / ml at the rate of 8ml per hour via a multiperforated catheter with connector after bolus of 20 ml
  Arms: intrathecal morphine

SUMMARY:
Analgesia in liver surgery is a challenge, postoperative coagulopathy risk raises fears an epidural haematoma formation following the epidural analgesia, "gold standard" in major abdominal surgery. The spinal analgesia and/or continuous wound infiltration of local anesthetics constitute so an alternative.

The study will compare the continuous infiltration of local anesthetics and rachianalgesia in terms of decreased postoperative morphine consumption and incidences of chronic postoperative pain at 3 and 6 months after hepatic surgery compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Surgery of hepatic resection by first under costal.
* Patient classified ASA 1 to 3.
* Information, signed and informed consent

Exclusion Criteria:

* Patients classified ASA 4 or 5.
* Allergy or intolerance to any of the products used in the protocol.
* Emergency surgery, palliative surgery, surgical recovery.
* History of chronic pain requiring the regular use of analgesics, especially opioids.
* History of drug misuse.
* Inability to understand and / or use the patient's self-controlled morphine pump.
* Known history of psychiatric disorders or current psychotropic treatment (excluding benzodiazepine monotherapy)
* Additive behavior with respect to alcohol or non-weaned psychodysleptic substances
* Pregnant Woman or Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2015-05-20 (Actual); Primary Completion 2019-05-25 (Actual); Study Completion 2019-05-25 (Actual)

PRIMARY OUTCOMES:
Morphine Consumption | During the first 24 hours post operative
  Morphine consumption is measured all 3 hours during the first 24 hours post operative

SECONDARY OUTCOMES:
Morphine Consumption | During the 48 hours post operative
  Morphine consumption is measured all 3 hours during the 48 hours post operative
Evaluation of postoperative pain intensity at rest | All 3 hours during the 48 postoperative hours
  The postoperative pain intensity is measured by Visual Analog Scale at rest
Evaluation of postoperative pain intensity after activity | All 3 hours during the 48 postoperative hours
  The postoperative pain intensity is measured by Visual Analog Scale after activity
Electric nociception threshold measured by PainMatcher | At the exit of Post Anesthesia Care Unit
  The Electric nociception threshold is measured by PainMatcher (CefarCompex®)
Electric nociception threshold measured by PainMatcher | At 24 hours post operative
  The Electric nociception threshold is measured by PainMatcher (CefarCompex®)
Electric nociception threshold measured by PainMatcher | At 48 hours post operative
  The Electric nociception threshold is measured by PainMatcher (CefarCompex®)
Number of patient with a chronic pain after liver surgery, measured by Questionnaire Douleur de Saint-Antoine (QDSA) | At 3 months after surgery
  Evaluation with validated score for chronic and neuropathic pains (QDSA is the French translation of the MPQ "Mac Gill bread questionary")
Number of patient with a chronic pain after liver surgery, measured by Questionnaire Douleur de Saint-Antoine (QDSA) | At 6 months after surgery
  Evaluation with validated score for chronic and neuropathic pains (QDSA is the French translation of the MPQ "Mac Gill bread questionary")
Number of patient with a chronic pain after liver surgery, measured by Neuropathic Pain Symptom Inventory (NPSI) | At 3 months after surgery
  Evaluation with validated score for chronic and neuropathic pains (NPSI)
Number of patient with a chronic pain after liver surgery, measured by Neuropathic Pain Symptom Inventory (NPSI), | At 6 months after surgery
  Evaluation with validated score for chronic and neuropathic pains (NPSI)
Number of patient with a chronic pain after liver surgery, measured by Neuropathic pain diagnostic questionnaire (DN2), | At 3 months after surgery
  Evaluation with validated score for chronic and neuropathic pains (DN2)
Number of patient with a chronic pain after liver surgery, measured by Neuropathic pain diagnostic questionnaire (DN2), | At 6 months after surgery
  Evaluation with validated score for chronic and neuropathic pains (DN2)
Area peri-incisional hyperalgesia | At 48 hours post operative
  The Surface of the cutaneous Area peri-incisional hyperalgesia is measured by Von frey's Filament.
Number of nausea and/or vomiting episodes | At 24 hours after surgery
  Measured by collection of episodes of nausea and/or vomiting and consumption of anti-emetics
Number of nausea and/or vomiting episodes | At 48 hours after surgery
  Measured by collection of episodes of nausea and/or vomiting and consumption of anti-emetics
Number of nausea and/or vomiting episodes | At 72 hours after surgery
  Measured by collection of episodes of nausea and/or vomiting and consumption of anti-emetics
Number of patient with side effect of morphine consumption | Up to 72 hours after surgery
  Respiratory Depression, Urinary retention, Prurit
Time physiological function recovery | Up to the end of hospital stay, an average 10 days
  Nasogastric tube withdrawal time, Transit recovery, Ability to drink, to eat, to urinate, to walk
Length of hospital stay in intensive care unit | Up to the end of hospital stay,an average 10 days
Length of hospital stay | Up to the end of hospital stay , an average 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Lebuffe, MD, PhD, Principal Investigator — CHRU de Lille
Locations (1):
- CHRU , Hôpital Claude Huriez, Lille, France

REFERENCES:
- [Result] Rousseleau D, Plane B, Labreuche J, Pierache A, El Amine Y, Ethgen S, Wattier JM, Cirenei C, Boleslawski E, Lebuffe G. Comparison of catheter wound infusion, intrathecal morphine, and intravenous analgesia for postoperative pain management in open liver resection: randomized clinical trial. BJS Open. 2025 Jul 1;9(4):zraf074. doi: 10.1093/bjsopen/zraf074. PMID 40662757